CLINICAL TRIAL: NCT03029221
Title: Local Evaluation of Real Relationships
Status: Completed | Type: Observational
Sponsor: Children's Aid Society in Clearfield County (Other)
Collaborators: By The Numbers Data Analysis & Statistical Solutions (Unknown)
Responsible Party: Sponsor
Other Study IDs: 90FM0104-01-01
Record Dates: First submitted 2017-01-16; First posted 2017-01-24 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Family Relationships; Parent-Child Relationships

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Marriage & Relationship Ed Skills-Couples: This group will receive the PREP 8.0 curriculum developed by PREP. In Years 2-5, 4 7-week class series will be held each year in Clearfield and Centre Counties (PA); 32 adults will be served each year. In Year 1, 8 adults will be served. Couples will receive 11 hours of curriculum instruction. This group will also receive two 30-minute presentations on available financial management, and job and career advancement services through two partnering organizations (CareerLink and Central PA Community Action, Inc.). Participants will also have access to optional parenting skills training provided by CAS (i.e., Triple P - Positive parenting Program). Referrals to community agencies based on individual/family needs will be provided by participant's case managers, as needed.
  Interventions: Other: PREP 8.0 curriculum developed by PREP
- Marriage & Relationship Ed Skills-Individuals: This group will receive the Within My Reach curriculum developed by PREP. In Years 2-5, 4 9-week class series will be held each year in Clearfield and Centre Counties (PA); 32 adults will be served each year. In Year 1, 8 adults will be served. Participants will receive 15 hours of curriculum instruction. This group will also receive two 30-minute presentations on available financial management, and job and career advancement services through two partnering organizations (CareerLink and Central PA Community Action, Inc.). Participants will also have access to optional parenting skills training provided by CAS (i.e., Triple P - Positive parenting Program). Referrals to community agencies based on individual/family needs will be provided by participant's case managers, as needed.
  Interventions: Other: Within My Reach curriculum developed by PREP
- Pre-Marital Ed and Marriage Skills: This group will receive healthy marriage and relationship education to pre-marital couples using Within Our Reach 8 Hours curriculum developed by PREP. In Years 2-5, 9 10-hour weekend workshops will be held each year in nine central PA counties; 72 adults will be served each year. In Year 1, 24 adults will be served.
  Interventions: Other: Within Our Reach 8 Hours curriculum
- Marriage Enhancement and Marriage Skills: This group will receive healthy marriage and relationship education to married couples using Within Our Reach 8 Hours curriculum developed by PREP. In Years 2-5, 9 12-hour weekend workshops will be held each year in nine central PA counties; 174 adults will be served each year. In Year 1, 60 adults will be served.
  Interventions: Other: Within Our Reach 8 Hours curriculum

INTERVENTIONS:
Other: PREP 8.0 curriculum developed by PREP — healthy marriage and relationship education
  Groups: Marriage & Relationship Ed Skills-Couples
Other: Within My Reach curriculum developed by PREP — healthy marriage and relationship education
  Groups: Marriage & Relationship Ed Skills-Individuals
Other: Within Our Reach 8 Hours curriculum — healthy marriage and relationship education
  Groups: Marriage Enhancement and Marriage Skills; Pre-Marital Ed and Marriage Skills

SUMMARY:
This project evaluates Real Relationships, a program provided by the Children's Aid Society (CAS) in Clearfield County, and funded through the DHHS Healthy Marriage (and Responsible Fatherhood) program. Research questions focus on recruitment and retention of participants, and short- and long-term participant outcomes associated with different formats for offering the program.

DETAILED DESCRIPTION:
Only adult participants living in the community are included in the local evaluation. Three research questions are examined in detail by the local evaluation. First, what recruitment strategies are most effective in the rural service area of Real Relationships? The answers to this research question will increase the CAS's and the funder's understanding of recruitment in rural areas. Secondly, what are barriers to Real Relationships class/workshop attendance for adults who enrolled but did not participate in any workshops? Again, answers to this research question will increase CAS's and the funder's understanding of barriers to retention (from the point of entry into the program to when participation begins), particularly in rural areas. A better understanding of barriers at this point of the enrollment process can be used to develop programming that helps to avoid these barriers, and the development of programming aimed at reaching populations that have been missed due to specific barriers. Third, how do short- and long-term outcomes for participants who complete their Real Relationships class/workshop differ by the format of the class/workshop format (i.e., weekend workshop, multi-week classes)? The answers to this research question will increase CAS's and the funder's understanding of programming in this field by adding to the knowledge base regarding the most effective formats for achieving the outcomes relevant to the goals of Real Relationships. Results will also speak to the importance of other activities, such as case management and parenting classes, for achieving desired outcomes.

ELIGIBILITY:
Inclusion Criteria:

* living in the community

Exclusion Criteria:

* living in an institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who participate in Children's Aid Society's Real Relationships program who live in the coimmunity
Sampling Method: Non-Probability Sample
Enrollment: 1119 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Work on Serious Disagreement at Post-Survey | Pre-Survey and Post-Survey, which would range from 30 days to 10 weeks
  nFORM Question on Pre/Post Survey, & Follow-up Survey: when have serious disagreement with spouse, worked on it together to find a resolution
Change from Post-Survey in Work on Serious Disagreement at Follow-up Survey | Post-Survey and Follow-up Survey, up to 4 months
  nFORM Question on Pre/Post Survey, & Follow-up Survey: when have serious disagreement with spouse, worked on it together to find a resolution
Change from Baseline in Spending Time with Child at Post-Survey | Pre-Survey and Post-Survey, which would range from 30 days to 10 weeks
  nFORM Question on Pre/Post Survey, & Follow-up Survey: frequency of spending time with a child doing things that he/she likes to do
Change from Post-Survey in Spending Time with Child at Follow-up | Post-Survey and Follow-up Survey, up to 4 months
  nFORM Question on Pre/Post Survey, & Follow-up Survey: frequency of spending time with a child doing things that he/she likes to do
Change from Baseline in Use of Written Budget at Post-Survey | Pre-Survey and Post-Survey, which would range from 30 days to 10 weeks
  nFORM Question on Pre/Post Survey, & Follow-up Survey: use a written budget to plan spending
Change from Post-Survey in Use of Written Budget at Follow-up Survey | Post-Survey and Follow-up Survey, up to 4 months
  nFORM Question on Pre/Post Survey, & Follow-up Survey: use a written budget to plan spending

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Floro, Study Director — Children's Aid Society in Clearfield County
Locations (1):
- Children's Aid Society in Clearfield County, Clearfield, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No